CLINICAL TRIAL: NCT03361709
Title: The Effect of Intracameral Injection of Dexamethasone After Phacoemulsification in Diabetic Patients on Corneal Endothelial Cell Density
Brief Title: Effect of Intracameral Dexamethasone After Phacoemulsification in Diabetics on Corneal Endothelial Cell Density
Acronym: DIABEDEX
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Inability to perform the study at present time.
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ayman Gehad Elnahry, Clinical Demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CU201712
Record Dates: First submitted 2017-11-29; First posted 2017-12-05 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus; Corneal Endothelial Cell Loss; Dexamethasone Adverse Reaction; Corneal Endothelial Decompensation
MeSH Terms: conditions — Diabetes Mellitus; Corneal Endothelial Cell Loss | interventions — Dexamethasone; Calcium Dobesilate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone group (Active Comparator): Dexamethasone injected at conclusion of Phacoemulsification
  Interventions: Drug: Dexamethasone
- Non-dexamethasone group (Placebo Comparator): No dexamethasone will be injected at the conclusion of Phacoemulsification
  Interventions: Drug: Saline Solutions, Intraocular

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be injected intracamerally at the conclusion of Phacoemulsification
  Other Names: Decadron
  Arms: Dexamethasone group
Drug: Saline Solutions, Intraocular — Only saline will be injected intracamerally at conclusion of Phacoemulsification
  Arms: Non-dexamethasone group

SUMMARY:
The prevalence of diabetes mellitus (DM) is rapidly growing worldwide. One major concern with diabetes mellitus is how it may affect vision in different ways; including the increased risk of developing cataract. Several studies have found an association between diabetes mellitus and the development of cataract. In patients with DM, cataract progression is also faster and occurs at a younger age.5 While results for modern cataract surgery are satisfactory, cataract surgery in diabetic patients carries a higher risk of peri and post-operative complications than in non-diabetic patients. Several studies have shown that the corneal endothelial count of diabetic patients is decreased, with more damage occurring to corneal endothelial cells following phacoemulsification in diabetics than in non-diabetics. This is presumed to be due to increased vulnerability of corneal endothelial cells in diabetics and a delay in the repair process.

Administration of topical corticosteroids is the main method to control post-operative inflammation after phacoemulsification, however many studies have also proved the safety and efficacy of intracameral corticosteroids to control inflammation post-operatively. While intracameral triamcinolone is effective in controlling post-operative inflammation, elevation of intraocular pressure is a main concern.

Dexamethasone has been found to be effective in controlling post-operative inflammation with no effect on intraocular pressure. This may be due to its rapid turnover and short half-life. No studies however have been performed to evaluate the safety and benefit of intracameral injection of dexamethasone following phacoemulsification in diabetic patients. In the present study, investigators aim to evaluate this and determine its effect on the post-operative corneal endothelial cell density and corneal thickness.

DETAILED DESCRIPTION:
This is a prospective interventional randomized controlled cohort study to determine the safety and benefit of intracameral dexamethasone injection at the conclusion of phacoemulsification in diabetic patients with cataract.

All patients will undergo full ophthalmological examination including best corrected visual acuity (BCVA), intraocular pressure (IOP), anterior segment examination and fundus examination. History and control of diabetes mellitus will be recorded. Patients ≥ 40 years old with a visually significant cataract, who are known to be diabetic for more than 10 years and are free of exclusion criteria will be included in our study.

In addition to routine pre-operative cataract evaluation and investigations, patients will also undergo non-contact Specular Microscopy (Konan Medical, Inc., Hyogo, Japan) to record the pre-operative corneal endothelial cell density in the central cornea, as well as anterior-segment optical coherence tomography (AS-OCT, Optovue Inc., Fremont, CA, USA) to record pre-operative central corneal thickness (CCT).

Standard phacoemulsification will be performed using the Infiniti machine (Alcon, Fort Worth, Texas, USA) with the stop and chop technique, and 0.2 mg of dexamethasone in 0.05 ml will be injected intracamerally at the conclusion of surgery in half of the study eyes, assigned using a randomization method.

Post-operative examination will include BCVA, IOP measurement and level of anterior segment inflammation on days 1,7 and 30 of follow up. Specular microscopy and AS-OCT will be performed at day 30 of follow up. Ophthalmologist performing examinations and investigations will be masked to whether dexamethasone was injected or not to avoid bias.

The difference in mean corneal endothelial cell density before and after phacoemulsification will be compared between both groups. The difference in CCT, post-operative inflammation and IOP will also be compared between both groups.

All statistical analyses will be done using IBM SPSS v20.0 statistical software (IBM Corporation, NY, USA). Descriptive statistics will be calculated, and the data will be summarized as mean ± SD for numerical data, and as frequencies and percentages for categorical data. When the p-value is < 0.05 this will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 years old
* Type 1 or Type 2 diabetes duration ≥ 10 years
* Visually significant cataract

Exclusion Criteria:

* Dense central corneal opacities as dense nebulae and stromal dystrophies.
* Pre-operative endothelial cell count less than 1500 cell/mm2
* Fuchs dystrophy
* Associated ocular conditions that could affect endothelial cell count as glaucoma and uveitis
* Previous intraocular surgeries

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in corneal endothelial cell density before and after phacoemulsification | 1 month
  This will be assessed using specular microscopy

SECONDARY OUTCOMES:
Central corneal thickness | 1 month
  Using specular microscopy
Intraocular inflammation | 1 month
  Assessed clinically 1,7 and 30 days after operation
Intraocular pressure | 1 month
  Assessed clinically 1,7 and 30 days after operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Dahab, MD, Study Director — Cairo University; Ahmed A Abdel Azim, MD, Study Director — Cairo University; Shaimaa A Arfeen, MD, Study Director — Cairo University; Ayman GA Elnahry, Msc, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No